CLINICAL TRIAL: NCT05395780
Title: An Open-label, Multi-center Phase II Clinical Study on MAX-40279-01 as Second or Later Lines of Treatment of Advanced Gastric Cancer or Gastroesophageal Junction Cancer
Brief Title: A Phase 2 Study to Evaluate the Safety and Efficacy of Max-40279-01 in Patients With Advanced Gastric Cancer or Gastroesophageal Junction Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maxinovel Pty., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MAX-40279-006
Record Dates: First submitted 2022-05-19; First posted 2022-05-27 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2021-11

CONDITIONS: Gastric Cancer; Gastroesophageal Junction Cancer
Keywords: Advanced/ gastric cancer/ gastroesophageal junction cancer.
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-dose MAX-40279 group (Experimental): High-dose MAX-40279 capsule group (10-15 subjects, 70 mg, BID, PO)
  Interventions: Drug: MAX-40279
- Low-dose MAX-40279 group (Experimental): Low-dose MAX-40279 capsule group (10-15 subjects, 50 mg, BID, PO)
  Interventions: Drug: MAX-40279

INTERVENTIONS:
Drug: MAX-40279 — MAX-40279 capsule will be administered orally
  Other Names: MAX-40279-01 capsule

SUMMARY:
This is a single-arm, multi-center phase II clinical study to Evaluate the Safety and Efficacy of Max-40279-01 in Patients With advanced gastric cancer or gastroesophageal junction cancer.

DETAILED DESCRIPTION:
This is a single-arm, multi-center phase II clinical study.

This study intends to enroll 20-30 subjects with advanced GC or GEJ adenocarcinoma on second or later lines of treatment (the tumor tissues of ≥ 50% of subjects will be tested by RNAseq, with FGOP2 TPM ≥ 9). Subjects will be randomly assigned to cohort 1 or 2 in a 1:1 ratio:

Cohort 1: High-dose MAX-40279 group (10-15 subjects, 70 mg, BID, PO) Cohort 2: Low-dose MAX-40279 group (10-15 subjects, 50 mg, BID, PO)

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation in the clinical study; full understanding of and fully informed of the study and signing of the informed consent form (ICF); being willing to follow and able to complete all trial procedures.
2. Age ≥ 18 years and ≤ 80 years, male or female.
3. Patients with histologically or cytologically confirmed advanced gastric adenocarcinoma (GC) or gastroesophageal junction (GEJ) adenocarcinoma on the second or later lines of treatment who failed at least the first line of standard treatment.
4. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1 point.
5. Presence of measurable lesions meeting RECIST 1.1 criteria.
6. Expected survival ≥ 12 weeks.
7. Before administration, patients must provide 5-8 unstained tumor tissue slides (samples taken within 12 months before the first dose) or fresh tissue specimens of ≥ 2 mm3.
8. Adequate organ and bone marrow functions as defined below (no treatment with blood transfusion, albumin, recombinant human thrombopoietin, or colony-stimulating factor (CSF) within 14 days before the first dose of the investigational drug).
9. The interval between the first dose of the investigational drug and previous major surgery, treatment with medical devices, or local radiotherapy (excluding palliative radiotherapy) should be at least 28 days; that for previous cytotoxic chemotherapy, endocrinotherapy, or treatment with biologicals should be at least 21 days; that for previous hormonotherapy or minor surgery should be at least 14 days; that for treatment with small-molecule targeted drugs should be at least 14 days or 5 half-lives, whichever is longer;
10. Female patients of childbearing age must undergo a serum pregnancy test within 7 days before administration of the investigational drug and the results should be negative, and they should be willing to take medically accepted, effective contraceptive measures (e.g., intrauterine device, contraceptives, or condoms) during the study period and within 3 months after the last dose of the investigational drug; male patients with female partners of childbearing age should have been surgically sterilized, or agree to implement effective contraceptive measures during the study period and within 3 months after the last dose of the investigational drug.

Exclusion Criteria:

1. Those who were diagnosed of any other malignancies within 3 years before the first dose, except for basal cell or squamous cell skin cancer or carcinoma in situ that has been adequately treated.
2. Known allergy to the investigational drug or any of its excipients.
3. Those with known Her-2 positive gastric adenocarcinoma or GEJ adenocarcinoma receiving no previous treatment of the target (e.g., Herceptin®) (those with PD can be enrolled after treatment with Herceptin®).
4. Known and uncontrolled or symptomatic active central nervous system (CNS) metastasis manifested as clinical symptoms, cerebral edema, spinal cord compression, carcinomatous meningitis, leptomeningeal disease, and/or progressive growth. History of CNS metastases or spinal cord compression; those who received definite treatment and showed stable clinical manifestations after 4-week discontinuation of anticonvulsants and steroids before the first dose of the investigational drug can be enrolled in the study.
5. Any previous treatment-induced toxicity that has not been relieved to normal or grade ≤ 1 (NCI CTCAE v5.0) before the first dose (except for alopecia, grade ≤ 2 fatigue, poor appetite, and peripheral neurotoxicity).
6. Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS), active hepatitis B (HbsAg positive or HbcAb positive and HBV DNA is greater than ULN), hepatitis C (hepatitis C antibodies are positive, and HCV-RNA is greater than the lower limit of detection for analytical method), or coinfection of hepatitis B and hepatitis C.
7. Those with serious comorbidities, including but not limited to: uncontrollable active infections, active peptic ulcers, and decompensated respiratory disorders.
8. Those who have clinical symptoms or signs of gastrointestinal tract obstruction before the first dose and require parenteral fluid replacement or nutrition. Patients with inflammatory bowel diseases or chronic diarrhea. Patients who underwent total gastrectomy.
9. Presence of following conditions within 6 months before the first dose: myocardial infarction, serious/unstable angina, NYHA class > II cardiac insufficiency, poorly controlled arrhythmia (including QTcF intervals of > 450 ms for males and > 470 ms for females, by Fridericia's formula), or symptomatic congestive cardiac failure.
10. Hypertension that cannot be effectively controlled by antihypertensive drugs (systolic blood pressure > 140 mmHg or diastolic blood pressure > 90 mmHg).
11. Known hereditary or acquired hemorrhage and thrombophilia, such as hemophilia, coagulopathy, thrombocytopenia, and hypersplenism.
12. Presence of significant hemoptysis or daily hemoptysis of up to half a teaspoon (2.5 mL) or more within 2 months before the first dose.
13. Presence of clinically significant hemorrhage symptoms (e.g., hemorrhage of digestive tract) or hemorrhagic tendency within 3 months before the first dose, or vasculitis.
14. Presence of arterial/venous thromboembolic events within 6 months before the first dose, such as cerebrovascular accident (including transient ischemic stroke, cerebral hemorrhage, and cerebral infarction), deep venous thromboembolism, and pulmonary embolism.
15. Those requiring long-term anticoagulant therapy with warfarin or heparin or long-term antiplatelet therapy (aspirin ≥ 300 mg/d or clopidogrel ≥ 75 mg/d) during the study period.
16. Pregnant and breastfeeding patients.
17. Patients with other serious physical or mental diseases or laboratory test abnormalities that may increase the risks for participation in the study or interference with the study results, and patients who are deemed unsuitable to participate in the study as assessed by investigators.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Through study completion, an average of 1 year

SECONDARY OUTCOMES:
Progression free survival (PFS) | Through study completion, an average of 1 year
Duration of response (DoR) | Through study completion, an average of 1 year
Disease control rate (DCR) | Through study completion, an average of 1 year
Overall survival (OS) | Through study completion, an average of 1 year
Incidence and severity of adverse events (AEs) and serious adverse events (SAEs) and abnormalities in vital signs,electrocardiogram (ECG), and laboratory tests | Through study completion, an average of 1 year
Cmax | Through study completion, an average of 1 year
  Maximum plasma drug concentration of Max-40279
Tmax | Through study completion, an average of 1 year
  Time to maximum plasma concentration of Max-40279 Time to maximum plasma concentration of Max-40279 Time to maximum plasma concentration of Max-40279 Time to maximum plasma concentration of Max-40279
AUC | Through study completion, an average of 1 year
  Area under the time-concentration curve of Max-40279
Correlation between expression level and mutation of FGFR1OP2-related proteins and efficacy | Through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jingsu, China